CLINICAL TRIAL: NCT06826300
Title: Analysis of Muscle Strength and Stiffness and the Effect of Manual Therapy on the Time Travel Speed of Kart Drivers
Brief Title: Application of Elbow Manipulation in Archers
Acronym: Manual Therapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KB/519/2024
Record Dates: First submitted 2025-01-20; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Health
Keywords: go-kart drivers; muscle fatigue; recovery; manipulation
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assessment of the impact of acute manipulation effects on the strength and stiffness of selected mus (Experimental): This technique involves a low-amplitude, high-velocity push on the shoulder and elbow joints with an additional two-second tension
  Interventions: Other: Manual therapy; Other: Placebo

INTERVENTIONS:
Other: Manual therapy — This technique involves a low-amplitude, high-velocity push on the shoulder and elbow joints with an additional two-second tension
Other: Placebo — Performing manipulations without a two-second preliminary tension of the joint capsule in the shoulder and elbow joints.

SUMMARY:
The aim of this study was to: (i) assess the impact of maximal muscle strength and stiffness on EMG and Myoton parameters for selected upper limb muscles; and (ii) assess how manipulation of the initial 2-s tension phase, in particular involving muscle stretching, affects these EMG and Myoton parameters during karting training.

DETAILED DESCRIPTION:
EMG and Myoton measurements will be performed on selected muscles of the shoulder joint and forearm during karting drivers' training, initially at the beginning, after the athletes perform their first 8-minute run, after manipulation and after another 8-minute run.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons aged 18,
* A license to drive a kart,
* A competitor who regularly competes in the league,
* Expressing informed consent to participate in the study and undertakes to comply with the regulations on the track and wear a helmet.

Exclusion Criteria:

* Lack of volunteer consent,
* Previous upper, lower limb and spine surgeries,
* Other upper limb injuries in the last 6 months,
* Pain limiting participation in the study,
* Neurological diseases,
* Connective tissue diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-09 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of MVC. | The study will be conducted 4 times during one training session (before the intervention, after the intervention, after race 1 and after race 2). Each isometric muscle test lasts 3 seconds.
  Muscle EMG is an assessment of electrical characteristics during the test, the electrical source of which is the muscle membrane potential, and measured in μV.
2 Assessment of MVC. | The study will be conducted 4 times during one training session (before the intervention, after the intervention, after race 1 and after race 2).Each isometric muscle test lasts 3 seconds.
  Muscle EMG is an assessment of electrical characteristics during the test, which is measured by the repetition frequency of muscle motor unit discharges, which is measured in Hz, at the same time of the test.
3. Muscle stiffness | The study will be conducted 4 times during one training session (before the intervention, after the intervention, after race 1 and after race 2). Each Myoton application lasts 1 sec for one point.
  Muscle stiffness - characteristic resistance to physical contraction, which deforms initially forming. Stiffness (N/m) was calculated as S = amax.mprobe/Δl.

CONTACTS AND LOCATIONS:
Locations (1):
- Go-Kart Track E1GOKARTS, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No
Once the study is complete, the results will be sent to the researcher who will analyze the data.